CLINICAL TRIAL: NCT04780815
Title: An Exploratory PET-study of Deposition, Disposition and Brain Uptake of [11C]Nicotine After Inhalation of 2 Nicotine Formulations Via the myBluTM E-cigarette in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial Brands PLC (Industry)
Collaborators: Nerudia Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NER 03/001
Record Dates: First submitted 2021-02-23; First posted 2021-03-04 (Actual); Results first posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- myBluTM Formulation 1 Oral cavity and lungs (Experimental): This group was used for measuring oral cavity and lungs endpoints after administration of Formulation 1
  Interventions: Other: myBluTM Formulation 1
- myBluTM Formulation 2 Oral cavity and lungs (Experimental): This group was used for measuring oral cavity and lungs endpoints after administration of Formulation 2
  Interventions: Other: myBluTM Formulation 2
- myBluTM Formulation 1 Brain (Experimental): This group was used for measuring brain endpoints after administration of Formulation 1
  Interventions: Other: myBluTM Formulation 1
- myBluTM Formulation 2 Brain (Experimental): This group was used for measuring brain endpoints after administration of Formulation 2
  Interventions: Other: myBluTM Formulation 2

INTERVENTIONS:
Other: myBluTM Formulation 1 — 1-2 puffs of each 3-5 seconds duration taken from myBluTM with Formulation 1, with inhalation of the vapour into the lungs
  Arms: myBluTM Formulation 1 Brain; myBluTM Formulation 1 Oral cavity and lungs
Other: myBluTM Formulation 2 — 1-2 puffs of each 3-5 seconds duration taken from myBluTM with Formulation 2, with inhalation of the vapour into the lungs
  Arms: myBluTM Formulation 2 Brain; myBluTM Formulation 2 Oral cavity and lungs

SUMMARY:
This is a single-center, exploratory positron emission tomography (PET) study of deposition, disposition and brain uptake [11C]nicotine when given to smokers as two different formulations via mybluTM e-cigarette system.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥18.0 and ≤ 30.0 kg/m2
* Habitual daily cigarette smoker
* Women have to be of non-child bearing potential

Exclusion Criteria:

* History of any clinically significant disease
* Relevant concomitant medication
* Any clinically significant condition
* Malignancy within the past 5 years
* Positif for HIV, hepatitis B or C
* Untreated hypertension
* Previous participation to a PET-study or other nuclide medical study
* Previous exposure to significant radiation
* Negative results of the modified Allen test on both arms at screening
* Alcohol or drug abuse

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PET Centre, Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | myBluTM Formulation 1 Oral Cavity and Lungs | myBluTM Formulation 2 Oral Cavity and Lungs | myBluTM Formulation 1 Brain | myBluTM Formulation 2 Brain
Started | 6 | 5 | 3 | 2
Completed | 6 | 5 | 3 | 1
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | myBluTM Formulation 1 Oral Cavity and Lungs | myBluTM Formulation 2 Oral Cavity and Lungs | myBluTM Formulation 1 Brain | myBluTM Formulation 2 Brain | Total
Number analyzed (Participants) | 6 | 5 | 3 | 1 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (2.8) | 54.2 (3.1) | 61.3 (5.5) | 54.0 (0.0) | 57.8 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 1 | 12
  Male | 2 | 1 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 5 | 3 | 1 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Lung PET
Description: Peak accumulation of [11C]nicotine deposited in the lung during 40 minutes after product administration, using dynamic PET Digital Imaging and Communications in Medicine (DICOM) images over the lungs
Time Frame: 40 minutes
Measure: Mean (Standard Deviation); unit: Percentage of nicotine
Arm/Group | myBluTM Formulation 1 Oral Cavity and Lungs | myBluTM Formulation 2 Oral Cavity and Lungs
Number analyzed (Participants) | 4 | 5
Percentage of nicotine | 35.5 (9.1) | 31.0 (9.6)

2. Primary Outcome: Oral Cavity PET
Description: Peak accumulation of nicotine deposited in the oral cavity during 40 minutes after product administration, using dynamic PET Digital Imaging and Communications in Medicine (DICOM) images over the oral cavity
Time Frame: 40 minutes
Measure: Mean (Standard Deviation); unit: Percentage of nicotine
Arm/Group | myBluTM Formulation 1 Oral Cavity and Lungs | myBluTM Formulation 2 Oral Cavity and Lungs
Number analyzed (Participants) | 5 | 5
Percentage of nicotine | 9.26 (2.44) | 1.52 (1.39)

3. Primary Outcome: Brain PET
Description: Peak accumulation of nicotine deposited in the brain during 30 minutes after product administration, using dynamic PET Digital Imaging and Communications in Medicine (DICOM) images over the brain
Time Frame: 30 minutes
Population: Four subjects underwent a brain [11C]nicotine PET/CT scan, but the tracer inhalation failed for two of the subjects. Consequently, only two [11C]nicotine scans could be used for evaluation, one after inhalation of Formulation 1 and one after inhalation of Formulation 2.
Measure: Number; unit: Percentage of nicotine
Arm/Group | myBluTM Formulation 1 Brain | myBluTM Formulation 2 Brain
Number analyzed (Participants) | 1 | 1
Percentage of nicotine | 4.50 | 5.14

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | myBluTM Formulation 1 Oral Cavity and Lungs | myBluTM Formulation 2 Oral Cavity and Lungs | myBluTM Formulation 1 Brain | myBluTM Formulation 2 Brain
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/6 | 1/5 | 2/3 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | myBluTM Formulation 1 Oral Cavity and Lungs (N=6) | myBluTM Formulation 2 Oral Cavity and Lungs (N=5) | myBluTM Formulation 1 Brain (N=3) | myBluTM Formulation 2 Brain (N=1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0
Catheter site hypo-aesthesia (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT04780815/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT04780815/SAP_001.pdf